CLINICAL TRIAL: NCT02086357
Title: Investigation of Ultrasound Elastographic Techniques in Soft Tissue Pathology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RD13/10834; 14845 (Other: UKCRN)
Record Dates: First submitted 2014-01-23; First posted 2014-03-13 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Tissue Pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- SWUE
  Interventions: Procedure: SWUE

INTERVENTIONS:
Procedure: SWUE

SUMMARY:
Ultrasound (US)tissue elastography has recently been found to have a number of clinical applications in the assessment of soft tissue disease for example, in breast and thyroid pathology. There are few current studies exploring its use in musculoskeletal pathology, particularly a new technique called sheer wave ultrasound elastography (SWUE).

Magnetic Resonance (MR) elastography has shown wide reaching applications in orthopaedics, sports medicine and rheumatology and SWUE may have the potential to also demonstrate clinical effectiveness in these areas.

Our aim is to explore the effectiveness of this technique in the assessment of musculoskeletal pathology.

Participants will be recruited through current referral protocols and would undergo an additional elastographic investigation in addition to their standard US examination. This investigation will be conducted within the musculoskeletal US department at Chapel Allerton Hospital by trained musculoskeletal specialists. The study will be conducted over a period of approximately 24 months with quarterly review during this time.

ELIGIBILITY:
Inclusion Criteria:

* Have clinical symptoms and signs of soft tissue pathology
* Be able to give consent
* Be over 16 years of age

Exclusion Criteria:

* Unable to give consent
* 16years of age or less
* Multifactorial soft tissue pathology

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Musculoskeletal US department at Chapel Allerton Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Clinical effectiveness of Sheer wave ultrasound elastography (SWUE) in the assessment of soft tissue pathology | Baseline to 24 months
  Ability of SWUE to accurately detect soft tissue pathology when compared with standard ultrasound techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom